CLINICAL TRIAL: NCT04491422
Title: Same-Day PrEP Initiation and Sexual Health for Transgender Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC REF 0105-2020
Record Dates: First submitted 2020-07-16; First posted 2020-07-29 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: HIV; PrEP; Transgender Women; Sexually Transmitted Diseases, Bacterial
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to either quarterly Integrated Next Steps Counseling (iNSC) using point-of-care (POC) urine tenofovir (TFV) levels [intervention arm] or standard adherence counseling without drug level feedback [control arm].
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Integrated Next Steps Counseling using poi (Active Comparator): At quarterly visits, intervention arm participants will receive iNSC Support Level 1 to address PrEP adherence and sexual health needs. Those with urine TFV levels <1000 ng/mL will receive iNSC Support Level 2, in which participant responses to two 7-item questionnaires on PrEP adherence and sexual health will guide problem solving on improved dosing.
  Interventions: Combination Product: Integrated Next Steps Counseling with Real-Time Drug Level Feedback
- Standard adherence counseling (No Intervention): Control arm participants will receive standard adherence counseling.

INTERVENTIONS:
Combination Product: Integrated Next Steps Counseling with Real-Time Drug Level Feedback — Integrated next steps counseling with real-time drug level feedback using point-of-care urine tenofovir testing at quarterly visits
  Arms: Integrated Next Steps Counseling using poi

SUMMARY:
Transgender women (trans women; assigned male sex at birth but identify as female) are at high risk for HIV infection, and are an important, under-researched population in sub-Saharan Africa. Trans women have a 13 times greater risk of acquiring HIV than adults aged 15-49 years in the general population, and in Africa, trans women have nearly twice the HIV prevalence (25%) of men who have sex with men [MSM] (14%). Oral pre-exposure prophylaxis (PrEP) is an effective prevention tool that could change the trajectory of the HIV epidemic among the 25 million trans women globally, yet its use has been suboptimal in this vulnerable population. Same-day PrEP initiation is feasible and acceptable and improves retention in PrEP care in resource-rich settings. Same-day initiation of emtricitabine/tenofovir alafenamide (F/TAF), a new PrEP regimen, has not to our knowledge previously been evaluated as PrEP in African trans women. F/TAF is potentially more efficacious and safer than emtricitabine/tenofovir disoproxil fumarate (F/TDF) as shown in the recent DISCOVER trial. However, concerns about drug-drug interactions between feminizing hormonal therapy (FHT) and PrEP are a key potential adherence barrier for trans women. While PrEP drugs do not lower FHT levels, FHT decreases plasma TFV and (emtricitabine) FTC levels. Little is known about FHT use among African trans women taking F/TAF or how concerns about F/TAF-FHT interactions may influence PrEP adherence. Moreover, interventions to support PrEP adherence in this population are needed. Feedback about PrEP use has been shown to potentially improve PrEP adherence among MSM but has not been utilized among trans women. Key knowledge gaps include: 1) whether same-day PrEP can be successfully implemented for African trans women, 2) the impact of drug-level feedback on PrEP adherence, and 3) how use of FHT may influence PrEP adherence.

To address these questions, this protocol describes a randomized trial to evaluate the feasibility and acceptability of same day initiation of F/TAF PrEP, evaluate impact of drug-level feedback on PrEP adherence and characterize PrEP persistence, and in-depth interviews to explore how self-care interventions for sexual health influence prevention choices among trans women and their sexual partners. This will be the first clinical trial, to our knowledge, to evaluate F/TAF as PrEP for HIV-negative trans women in sub-Saharan Africa.

DETAILED DESCRIPTION:
The overall goal of this study is to evaluate the feasibility and acceptability of same-day F/TAF initiation and characterize F/TAF persistence among trans women taking PrEP. This research will be conducted at the Infectious Diseases Institute, Makerere University in Kampala, Uganda and consists of 3 complementary aims. In Aims 1 and 2, the investigators will assess the feasibility and acceptability of same-day F/TAF initiation and characterize PrEP persistence. In Aim 3, the investigators will use qualitative methods to explore how self-care interventions for sexual health influence prevention choices among trans women and their sexual partners. Study subjects will be accrued using respondent driven sampling (RDS) and enrolled at the study clinic where F/TAF will be initiated same day. Participants will be randomized in a 1:1 ratio to either the intervention arm (quarterly integrated next steps counseling [iNSC] using point-of-care [POC] urine tenofovir [TFV] levels) or the control arm (standard adherence counseling without drug level feedback). In Aim 3, the investigators will use qualitative methods to explore how self-care interventions for sexual health influence prevention choices among trans women and their sexual partners. The overall goal will be to assess whether POC urine testing and iNSC counseling increase PrEP uptake and persistence over 12 months. This study for trans women is guided by the cardinal ethical principles of justice, respect for persons and beneficence. The local trans community will be involved in study design and implementation.

Aim 1 : Evaluate the feasibility and acceptability of same-day F/TAF PrEP initiation among African trans women.

Approach: The investigators will recruit up to 200 trans women. All study participants who meet study eligibility criteria will be consented and enrolled at the study clinic. Randomization will occur through REDCap. Participants will start PrEP on the day of enrollment and receive F/TAF for 12 months. Free HIV and sexually transmitted infection (STI) testing and treatment will be provided to all participants.

Aim 2 : Characterize F/TAF persistence and test the impact of drug level feedback among African trans women taking PrEP.

Approach: Using a factorial design within the Aim 1 study, all F/TAF users will be randomized to real-time drug level feedback and adherence counseling using a POC urine TFV lateral-flow immunoassay versus standard counseling alone. Socio-behavioral surveys will assess potential factors influencing adherence, including gender dysphoria and FHT.

Aim 3 : Explore how self-care interventions for sexual health influence HIV/STI prevention choices among African trans women and their sexual partners.

Approach: To clarify how same-day PrEP initiation, FHT use and self-collection of samples (SCS) for STI testing may influence prevention choices, the investigators will conduct in-depth interviews with participants and their sexual partners to assess perceptions and experiences with same-day PrEP, real-time drug level feedback, use of FHT, SCS, and how self-care interventions could empower trans women to engage in prevention services.

Hypothesis: Same-day PrEP initiation will be a feasible and acceptable entryway into PrEP care among trans women.

ELIGIBILITY:
Inclusion Criteria:

* Report male sex assigned at birth but currently identify as female
* Age ≥18, or if 14-17 years, qualification as a mature or emancipated minor due to having a sexually transmitted infection or cater for own livelihood
* Report unprotected anal intercourse in the past 6 months
* Able and willing to provide written informed consent
* Possess a valid recruitment coupon
* HIV-uninfected based on negative HIV rapid tests at the enrollment visit

Exclusion Criteria:

* Currently enrolled in a biomedical HIV prevention study
* Any clinically significant or chronic medical condition that is considered progressive or in the opinion of the investigator would make the participant unsuitable for the study, including severe infections requiring treatment such as tuberculosis, alcohol or drug abuse, or mental illness which precludes provision of informed consent
* Not planning to remain in the geographic area for the duration of the study

Min Age: 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-identify as transgender women
Enrollment: 200 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of same-day initiation of F/TAF as PrEP as measured by participant engagement until the end of study | 12 months
  Proportion retained on PrEP at months 3, 6, 9 and 12
Acceptability of peer-delivered combination HIV prevention as measured by the System Usability Scale | 12 months
  System Usability Scale scores range from 0 to 100; higher scores mean better acceptability
Adoption of same-day PrEP initiation as measured by structured questionnaires | 12 months
  Proportion initiating same-day PrEP at enrollment
Fidelity to iNSC assessed through audio-recorded drug level feedback counseling sessions | 12 months
  Proportion of research nurses successfully implementing iNSC
PrEP persistence as measured by intracellular tenofovir diphosphate levels in dried blood spots at months 3, 6, 9, 12 | 12 months
  Proportion with tenofovir diphosphate levels >900 fmol per punch

SECONDARY OUTCOMES:
Sexual risk behaviors assessed through structured questionnaires | 12 months
  Proportion reporting unprotected sex, sexual frequency
STI incidence assessed through GeneXpert testing | 12 months
  Neisseria gonorrhoeae and Chlamydia trachomatis incidence

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mujugira, PhD, Principal Investigator — Infectious Diseases Institute
Locations (1):
- Infectious Diseases Institute Kasangati, Kampala, Uganda